CLINICAL TRIAL: NCT02407834
Title: Clinical Evaluation of an Experimental Solution Based on Ricinus Communis Compared to Sodium Hypochlorite for Denture Cleansing
Brief Title: Effectiveness of Hygiene Solutions on Denture Biofilm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Cláudia Helena Lovato da Silva, Cláudia Helena Lovato da Silva, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: mestradopt2013
Record Dates: First submitted 2015-02-09; First posted 2015-04-03 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Stomatitis
Keywords: Biofilms; Dentures; Denture Cleansers; Castor Oil; Stomatitis
MeSH Terms: conditions — Stomatitis | interventions — S 1 (combination); Sodium Hypochlorite; Epinephrine; Castor Oil; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- S1 - 0.25% sodium hypochlorite (Experimental): Brushing with specific brush and neutral soap, three times a day. After, immesion in 0.25% sodium hypochlorite during 20 minutes, once a day. This protocol was used during 7 days.
  Interventions: Other: S1
- S2 - 0.5% sodium hypochlorite (Experimental): Brushing with specific brush and neutral soap, three times a day. After, immesion in 0.5% sodium hypochlorite during 20 minutes, once a day.This protocol was used during 7 days.
  Interventions: Other: S2
- S3 - 10% Ricinus communis (Experimental): Brushing with specific brush and neutral soap, three times a day. After, immesion in 10% Ricinus communis solution during 20 minutes, once a day. This protocol was used during 7 days.
  Interventions: Other: S3
- S4 - saline solution (Placebo Comparator): Brushing with specific brush and neutral soap, three times a day. After, immesion in saline solution during 20 minutes, once a day. This protocol was used during 7 days.
  Interventions: Other: S4

INTERVENTIONS:
Other: S1 — Immersion in 0.25% sodium hypochlorite for 20 minutes, during 7 days.
  Other Names: 0.25% sodium hypochlorite
  Arms: S1 - 0.25% sodium hypochlorite
Other: S2 — Immersion in 0.5% sodium hypochlorite for 20 minutes, during 7 days.
  Other Names: 0.5% sodium hypochlorite
  Arms: S2 - 0.5% sodium hypochlorite
Other: S3 — Immersion in 10% Ricinus communis for 20 minutes, during 7 days.
  Other Names: 10% ricinus communis
  Arms: S3 - 10% Ricinus communis
Other: S4 — Immersion in Saline solution for 20 minutes, during 7 days.
  Other Names: saline solution
  Arms: S4 - saline solution

SUMMARY:
This clinical trial evaluated Ricinus communis and sodium hypochlorite solutions in different concentrations for denture cleanliness, regarding biofilm removal capacity, remission of atrophic chronic candidiasis, degree of patient satisfaction and antimicrobial action against specific microorganism. Sixty-four denture wearers with absence (n=40) or presence of Candidiasis (n=24) were selected and oriented to brush their dentures with a specific brush and neutral soap for 3 minutes, 3 times a day and immerse them, once a day, in hygiene solutions (0.25% sodium hypochlorite - S1 and 0.5% - S2, 10% R. communis - S3; Saline - S4: control) during 20 minutes, for 7 days. The solutions were used in a randomized, double blind and cross form with washout periods. To quantify biofilm with software ImageTool 3.0, the inner surface was disclosed (1% neutral red) and photographed at the end of each period. The Candidiasis remission was assessed by scores before and after the use of solutions. Patient satisfaction was assessed by questionnaire. Antimicrobial activity was determined by Colony Forming Units (CFU) counts of Streptococcus mutans, Candida spp., and gram-negative microorganisms. For collecting biofilm, internal surface of each maxillary complete denture was brushed with saline solution, and the biofilm suspension obtained. After serial dilutions (100 - 10-3), 50 uL aliquots were seeded in Petri dishes containing Mitis salivarius agar base, CHROMagar Candida® and MacConkey agar for detecting S. mutans, Candida spp., or gram-negative microorganisms, respectively. After incubation, colonies were counted, and values in CFU/mL were calculated. Biofilm removal was analyzed as a split-plot with two variation factors: inflammation and solutions. The candidiasis remission was analyzed after adjustment using multinomial logistic regression. Logistic regression analysis and compound symmetry was adopted for patient satisfaction. The antimicrobial action was analyzed with Friedman´s test. Antimicrobial action data were processed after transformation - log10 (CFU + 1) - and were analyzed by Friedman test (α = 0.05).

DETAILED DESCRIPTION:
Sixty-four denture wearers with (n=24) and without Candidiasis (n=40) were enrolled and instructed to brush and immerse their dentures in 4 different storage solutions (S1: 0.25% sodium hypochlorite; S2: 0.5% sodium hypochlorite; S3: 10% R. communis; and S4: Saline/Control). The interventions were randomly performed in a double blind and crossover format with washout periods. After 7 days of brushing and storage, the biofilm formed in the inner surfaces of dentures was disclosed and photographed to quantification. Candidiasis remission was assessed by scores and the patient satisfaction by a questionnaire. Antimicrobial activity of the solutions was determined by counting the Colony Forming Units (CFUs) of Streptococcus mutans, Candida spp., and gram-negative microorganisms. For collecting biofilm, each complete upper denture was placed in a Petri dish, its internal surface was brushed (Tek brush) with saline solution for 2 min, and the biofilm suspension was transferred to a test tube. After serial dilutions (100 - 10-3), 50 uL aliquots were seeded in Petri dishes containing Mitis salivarius agar base, CHROMagar Candida® and MacConkey agar for detecting S. mutans, Candida spp., or gram-negative microorganisms, respectively. After incubation, colonies were counted, and values in CFU/mL were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Edentulous that make regular use of dentures in acrylic resin for at least one year with the presence of biofilm.

Exclusion Criteria:

* Problems in adapting, reline, or repair fractures
* Patients with limited communication or collaboration as the following recommended protocol.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
biofilm removal capacity using Image Tool software | 7 days
antimicrobial action against specific microorganisms by Colony Forming Units counts | 7 days

SECONDARY OUTCOMES:
remission of atrophic chronic candidiasis using multinomial logistic regression analysis | 7 days
degree of patient satisfaction assessed by specific questionnaire | 7 days